CLINICAL TRIAL: NCT00606307
Title: A Phase IIA Study of the Histone-deacetylase Inhibitor ITF2357 in Patients With JAK-2 V617F Positive Chronic Myeloproliferative Diseases
Brief Title: Phase IIA Study of the HDAC Inhibitor ITF2357 in Patients With JAK-2 V617F Positive Chronic Myeloproliferative Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSC/07/2357/28
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Myeloproliferative Diseases
Keywords: polycythemia vera (PV); essential thrombocythemia (ET); myelofibrosis (MF)
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis | interventions — givinostat hydrochloride; givinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ITF2357 (Experimental): Initial dose of 50 mg b.i.d. that was subsequently escalated to 50 mg t.i.d in case of lack of significant toxicity.
  Interventions: Drug: ITF2357

INTERVENTIONS:
Drug: ITF2357 — 50 mg b.i.d. PO every day. More precisely, ITF2357 was supplied as 50 mg hard gelatine capsules for oral administration.
  Other Names: Givinostat

SUMMARY:
Primary Objective:

To evaluate efficacy and safety of ITF2357 in the treatment of patients with JAK2V617F positive myeloproliferative diseases [Polycythemia Vera (PV), Essential Thrombocytosis (ET), Myelofibrosis (MF)]. Efficacy was evaluated by ad hoc haematological and clinical criteria for PV and ET, and by internationally established response criteria (EUMNET criteria) for MF. Safety was evaluated by number of subjects experiencing an Adverse Event (AE), type, frequency, severity, timing and relatedness of AEs, including changes in vital signs and clinical laboratory results.

Secondary Objective:

To evaluate the JAK2 mutated allele burden by quantitative Real-Time Polymerase Chain Reaction (qRTPCR).

DETAILED DESCRIPTION:
This is a non-randomized, open-label, Phase IIA pilot study testing efficacy and safety of ITF2357 in a population of patients with JAK2V617F positive myeloproliferative diseases. All recruited patients received an initial dose of 50 mg b.i.d. of ITF2357 that was subsequently escalated to 50 mg t.i.d. in case of lack of significant toxicity. Treatment lasted up to a maximum of 24 cumulative weeks of drug administration. The study was carried out in Italy. Enrolled patients were subjects of both genders, with an established diagnosis of polycythemia vera (PV), essential thrombocythemia (ET) and myelofibrosis (MF) according to the revised WHO criteria.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Male or female, age ≥ 18 years
* Confirmed diagnosis of PV/ET/MF according to the revised World Health Organisation criteria
* JAK-2 V617F positivity
* In need of cytoreductive therapy when hydroxyurea is not indicated (e.g. young patients) or when refractoriness to the drug is documented

Exclusion Criteria:

* Active bacterial or fungal infection requiring antimicrobial treatment on Day 1
* Patients of childbearing potential without a negative pregnancy test prior to initiation of the study drug
* Pregnancy or lactation
* A marked baseline prolongation of QT/QTc interval (e.g. repeated demonstration of a QTc interval > 450 ms, according to Bazett's correction formula - see appendix G for the formula)
* The use of concomitant medications that prolong the QT/QTc interval (see appendix F for full list)
* Concomitant acute coronary syndromes; uncontrolled hypertension
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of any cardiac arrhythmia requiring medication (irrespective of its severity)
* A history of additional risk factors for Torsade de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* Active Epstein Barr Virus (EBV) infection (i.e. positive serology IgM)
* Known HIV infection
* Active hepatitis B and/or C infection
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk from treatment complications
* Eastern Cooperative Oncology Group (ECOG) performance status 3 or greater
* Platelets count <100x109/L within 14 days before enrolment
* Absolute neutrophil count <1.2x109/L within 14 days before enrolment
* Percentage of blast cells in peripheral blood >10% within 14 days before enrolment
* Serum creatinine >2xULN (Upper limit of normal)
* Total serum bilirubin >1.5xULN
* Serum AST (aspartate aminotransferase) / ALT (alanine aminotransferase) > 3xULN
* Interferon alpha within 14 days before enrolment
* Hydroxyurea within 14 days before enrolment
* Anagrelide within 7 days before enrolment
* Any other investigational drug within 28 days before enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: tiziano oldoni, MD, Study Director — Italfarmaco; Alessandro Rambaldi, MD, Principal Investigator — A.O. Ospedale Papa Giovanni XXIII
Locations (2):
- Italy (2):
  - Ospedali riuniti, Bergamo
  - IRCCS - Pol. San Matteo, Pavia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ITF2357
Started | 29
Completed | 18
Not Completed | 11
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — Disease progression | 6
Not completed — QTc prolongation | 1

BASELINE CHARACTERISTICS:
Arm/Group | ITF2357
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14.0
  Male | 15.0
Region of Enrollment [Number; unit: participants]
  Italy | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Objective Responses (Complete, Major, Moderate or Minor Responses), in Terms of Best Overall Response
Description: Patients with Objective Response were defined as those patients achieving a complete, major, moderate or minor (only for Myelofibrosis patients) response during the experimental treatment course.
  The "best response" is reported hereunder by intensity of response.
Time Frame: Every single week from week 1 to week 24 of treatment
Population: ITT population: all recruited patients who received study medication and for whom at least one on-study tumour evaluation is available.
Measure: Count of Participants; unit: Participants
Arm/Group | ITF2357
Number analyzed (Participants) | 29
Participants
  complete responders | 2
  major responders | 12
  moderate responders | 2
  minor responders | 1
  non responders | 12

2. Secondary Outcome: Change in JAK2 Mutated Allele Burden
Description: This outcome was assessed by quantitative real time Polymerase Chain Reaction (RT PCR).
  At each time point, the number of patients is the following:
  Screening: N=29 Week 12: N=20 Week 24: N=18 EOT: N=24. End of treatment corresponds to the last visit performed before treatment discontinuation.
Time Frame: At screening, at week 12, at week 24, at the end of treatment (EOT) visit
Population: Intent-to-treat population: all recruited patients who received study medication and for whom at least one on-study tumour evaluation is available.
Measure: Mean (Standard Deviation); unit: percentage of change in allele burden
Arm/Group | ITF2357
Number analyzed (Participants) | 29
percentage of change in allele burden
  screening | 54.0 (19.7)
  week 12: number analyzed (Participants) | 20
  week 12 | 49.4 (20.1)
  week 24: number analyzed (Participants) | 18
  week 24 | 47.1 (20.0)
  EOT: number analyzed (Participants) | 24
  EOT | 49.0 (21.5)

3. Secondary Outcome: Number of Subject Experiencing an Adverse Event
Description: An adverse event (AE) is any untoward occurrence in a patient or clinical investigation subject administered with a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  The adverse events must to be followed to the end of study (28 days after the last study drug intake).
  A serious AE (SAE) is defined as an untoward (unfavourable) medical occurrence that at any dose results in death, or is life-threatening or requires inpatient hospitalisation or prolongation of existing hospitalisation, or results in persistent or significant disability/incapacity or is a congenital anomaly/birth defect.
Time Frame: At weekly visits (Days 8, 15, 22, 36, 43, 50, 64, 71, 78, 99, 127, 155); At monthly visits (Days 29, 57, 85 113, 141,169); at end of treatment visit
Population: safety population: all recruited patients who received at least one dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | ITF2357
Number analyzed (Participants) | 29
Participants
  number of patients with AE | 29
  number of patients with serious AE | 3

ADVERSE EVENTS:
Time Frame: At weekly visits (Days 8, 15, 22, 36, 43, 50, 64, 71, 78, 99, 127, 155); At monthly visits (Days 29, 57, 85 113, 141,169); at three-monthly visit (Day 85)
Arm/Group | ITF2357
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 3/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITF2357 (N=29)
Cellulitis (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Melena (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITF2357 (N=29)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Cardiac disorders) | 3 (3)
Palpitation (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 18 (18)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Rectal Haemorrhage (Gastrointestinal disorders) | 2 (2)
Vomiting (General disorders) | 1 (1)
Asthenia (General disorders) | 9 (9)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Oedema peripheral (Hepatobiliary disorders) | 2 (2)
Pyrexia (Hepatobiliary disorders) | 8 (8)
Hypertransaminasaemia (Hepatobiliary disorders) | 2 (2)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 2 (2)
Cystitis escherichia (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Gastritis bacterial (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 5 (5)
Oral candidiasis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase (Investigations) | 1 (1)
Aspertate aminotransferase (Investigations) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 5 (5)
Weight decreased (Investigations) | 12 (12)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscoloskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Neurological symptom (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Renal and urinary disorders) | 1 (1)
sciatica (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Breast discomfort (Reproductive system and breast disorders) | 1 (1)
Gynaecomastia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Surgical and medical procedures) | 3 (3)
Rush (Surgical and medical procedures) | 2 (2)
Astringent therapy (Surgical and medical procedures) | 1 (1)
Angiopathy (Vascular disorders) | 1 (1)
Erythromelalgia (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Non reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No